CLINICAL TRIAL: NCT03029455
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Dose Escalation, and Bioavailability Study Evaluating the Safety and Pharmacokinetics of VX-659 in Healthy Subjects and in Subjects With Cystic Fibrosis
Brief Title: A Study to Evaluate Safety and Pharmacokinetics of VX-659 in Healthy Subjects and in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX16-659-001; 2016-003048-35 (EudraCT Number)
Record Dates: First submitted 2017-01-11; First posted 2017-01-24 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — VX-659; tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A: VX-659 or Matching Placebo (Experimental): Part A includes single-dose escalation.
  Interventions: Drug: VX-659; Drug: VX-659 Matching Placebo
- Part B: VX-659 or Matching Placebo (Experimental): Part B includes multiple-dose escalation.
  Interventions: Drug: VX-659; Drug: VX-659 Matching Placebo
- Part C: VX-659 in TC with TEZ/IVA or Matching Triple Placebo (Experimental): Part C includes multiple dose escalation of VX-659 administered in Triple Combination (TC).
  Interventions: Drug: VX-659; Drug: Tezacaftor; Drug: Ivacaftor; Drug: Triple Combination (TC) Matching Placebos
- Part D: VX-659 in TC with TEZ/IVA or Matching Triple Placebo (Experimental): Part D includes subjects with CF. Participants will receive TC or matching placebos.
  Interventions: Drug: VX-659; Drug: Tezacaftor; Drug: Ivacaftor; Drug: Triple Combination (TC) Matching Placebos

INTERVENTIONS:
Drug: VX-659
Drug: Tezacaftor
  Other Names: VX-661; TEZ
  Arms: Part C: VX-659 in TC with TEZ/IVA or Matching Triple Placebo; Part D: VX-659 in TC with TEZ/IVA or Matching Triple Placebo
Drug: Ivacaftor
  Other Names: VX-770; IVA
  Arms: Part C: VX-659 in TC with TEZ/IVA or Matching Triple Placebo; Part D: VX-659 in TC with TEZ/IVA or Matching Triple Placebo
Drug: VX-659 Matching Placebo
  Arms: Part A: VX-659 or Matching Placebo; Part B: VX-659 or Matching Placebo
Drug: Triple Combination (TC) Matching Placebos
  Arms: Part C: VX-659 in TC with TEZ/IVA or Matching Triple Placebo; Part D: VX-659 in TC with TEZ/IVA or Matching Triple Placebo

SUMMARY:
Evaluate the safety and tolerability of VX-659 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers: PARTS A, B, and C

* Males and Females of non-childbearing potential.
* Between the ages of 18 and 60 years inclusive
* Healthy, as defined per protocol.
* Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive
* Body weight >50 kg

CF Patients: PART D

* Body weight ≥35 kg.
* Males and Females of non-childbearing potential.
* Sweat chloride value ≥ 60 mmol/L at screening.
* Heterozygous for F508del and a minimal function CFTR mutation
* Forced expiratory volume in 1 second (FEV1) ≥40% and ≤90% of predicted at screening

Exclusion Criteria:

Healthy Volunteers: PARTS A, B, and C

* History of any illness or any clinical condition that in the opinion of the investigator might confound the results of the study or pose additional risk to the subject.
* Any condition possibly affecting drug absorption.
* History of febrile illness within 14 days before the first study drug dose.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency assessed at Screening.

CF Patients: PART D

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the subject.
* History of cirrhosis with portal hypertension.
* Risk factors for Torsade de Pointes.
* G6PD deficiency assessed at Screening.
* Abnormal Laboratory Values.
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* History of solid organ or hematological transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessments as determined by number of subjects with adverse events (AEs) and serious adverse events (SAEs) | from baseline up to Day 50

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of VX-659 and selected metabolites (μg/mL) | from baseline up to Day 18
Cmax of TEZ and selected metabolites (μg/mL) | from baseline up to Day 18
Cmax of IVA and selected metabolites (μg/mL) | from baseline up to Day 18
Area under the concentration versus time curve during a dosing interval (AUCtau) of VX-659 and selected metabolites (μg,h/mL) | from baseline up to Day 18
AUCtau of TEZ and selected metabolites (μg,h/mL) | from baseline up to Day 18
AUCtau of IVA and selected metabolites (μg,h/mL) | from baseline up to Day 18
Observed pre-dose concentration (Ctrough) of VX-659 and selected metabolites (μg/mL) | from baseline up to Day 18
Ctrough of TEZ and selected metabolites (μg/mL) | from baseline up to Day 18
Ctrough of IVA and selected metabolites (μg/mL) | from baseline up to Day 18

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Birmingham
  - Cambridge
  - Exeter
  - Glasgow
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Southampton

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Davies JC, Moskowitz SM, Brown C, Horsley A, Mall MA, McKone EF, Plant BJ, Prais D, Ramsey BW, Taylor-Cousar JL, Tullis E, Uluer A, McKee CM, Robertson S, Shilling RA, Simard C, Van Goor F, Waltz D, Xuan F, Young T, Rowe SM; VX16-659-101 Study Group. VX-659-Tezacaftor-Ivacaftor in Patients with Cystic Fibrosis and One or Two Phe508del Alleles. N Engl J Med. 2018 Oct 25;379(17):1599-1611. doi: 10.1056/NEJMoa1807119. Epub 2018 Oct 18. PMID 30334693